CLINICAL TRIAL: NCT03707145
Title: Effect of Online Support and Patient Empowerment on Functional Ability and Well-being in Older Adults: a Pilot Study
Brief Title: FrAilty Care and wEll-funcTion in Community Dwelling Older Adults
Acronym: FACET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aberystwyth University (Other)
Collaborators: EIT Health (Other)
Responsible Party: Principal Investigator, Marco Arkesteijn, Lecturer in Sport and Exercise Biomechanics, Aberystwyth University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 9526
Record Dates: First submitted 2018-09-06; First posted 2018-10-16 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-07

CONDITIONS: Frailty; Sarcopenia; Aging
Keywords: well-being; exercise; physical activity; nutrition; gait
MeSH Terms: conditions — Frailty; Sarcopenia; Motor Activity | interventions — Referral and Consultation; Diet; Exercise

STUDY DESIGN:
Intervention Model Description: Randomised; Interventional; Design type: Treatment, Complex Intervention, Physical, Rehabilitation
Who Masked: Participant
Masking Description: The participant is unaware of the other groups details. Assessor and investigator are not blinded due to the need for providing information to the participant about their group allocation in this pilot project
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Professional led with online support (Active Comparator): The consultation is led by the professional and lifestyle recommendations are based on ViviFrail recommendations and personal experience of the professional.
  The 12-week intervention includes access to an online monitoring platform. The online platform provides the lifestyle recommendations and consists of a diary of activities, examples of exercises, general advice and instructions for monitoring and self-assessment.
  Interventions: Behavioral: Consultation; Behavioral: Online Support
- Professional led without online support (Active Comparator): The consultation is led by the professional and lifestyle recommendations are based on ViviFrail recommendations and personal experience of the professional.
  There is no access to the online monitoring platform, and lifestyle recommendations were provided on paper to the participant.
  Interventions: Behavioral: Consultation
- Patient empowered with online support (Experimental): The consultation is led by the participant, and started with the questions 'What matters to you', and 'What are your goals'. The professional based the lifestyle recommendations based on these responses.
  The 12-week intervention includes access to an online monitoring platform. The online platform provides the lifestyle recommendations and consists of a diary of activities, examples of exercises, general advice and instructions for monitoring and self-assessment.
  Interventions: Behavioral: Consultation; Behavioral: Online Support; Behavioral: Empowered
- Patient empowered without online support (Active Comparator): The consultation is led by the participant, and started with the questions 'What matters to you', and 'What are your goals'. The professional based the lifestyle recommendations based on these responses.
  There is no access to the online monitoring platform, and lifestyle recommendations were provided on paper to the participant.
  Interventions: Behavioral: Consultation; Behavioral: Empowered

INTERVENTIONS:
Behavioral: Consultation — The consultation will provide advice (including a short written report) about promoting healthy lifestyles, tailored to the individual
  Other Names: Diet, exercise and physical activity advice
Behavioral: Online Support — The participant will have access to an online platform 'FACET', to monitor themselves periodically, obtain feedback about their functional ability, receive recommended diet, exercise and physical activity interventions and record the adherence to any intervention.
  Arms: Patient empowered with online support; Professional led with online support
Behavioral: Empowered — The participant will be actively encouraged to contribute to their own consultation and take co-ownership and responsibility for the action plan.
  Arms: Patient empowered with online support; Patient empowered without online support

SUMMARY:
This study is looking at whether older people could benefit from an online monitoring platform to support their individual ambitions to maintain or improve functional ability. It is hypothesized this will enable the individual to monitor themselves periodically, obtain feedback about their functional ability, receive recommended diet, exercise and physical activity interventions and record the adherence to any intervention. All information can be linked back to the health care professional for official support and intervene when a decline is noticed, in order to prevent frailty from developing. The aim of this study is to find out if providing more support and greater empowerment can help older people improve their functional ability by self-monitoring and personalised interventions.

DETAILED DESCRIPTION:
Participants will be individually randomised using randomisation service on a 1:1 allocation ratio to either group. There will be 4 groups, with differences in the consultation design and online support available.

Participant assessments consists of questionnaires and physical tasks completed during two visits at the university facilities. During the second visit, a one-hour consultation with a health care professional will take place to develop a twelve-week action plan to promote a healthier lifestyle.

Frailty status will be defined from the Fried frailty phenotype criteria. Exercise status will be based on current physical activity levels and the Short Physical Performance Battery score derived from the chair-stands, gait speed and balance assessments.

Participants in the experimental group will receive the assessment, and the consultation will aim to promote to empower them, plus access to the online support platform, termed 'FACET'.

Participants in the empowerment groups are provided with a structured booklet prior to the consultation to help the participant actively contribute to their own intervention programme, whereas in the other groups,the professional will lead the consultation.

Participants in the online support groups are provided with FACET, which will provide a diary of recommended activities to do, assessments to complete, as well as information about healthy lifestyles, diet and physical activity recommendations. Details on the recommended exercises and diet will be provided (including demonstrations and examples, also sourced from reputable websites) via FACET and will enable the participant to engage with them. The exercises require no special equipment and can be performed without professional supervision. Participants will be able to monitor themselves regularly and progress or amend recommendations to tailor their needs. Progress will also be monitored by the initial assessors and these can also amend the recommendations based on participant feedback. In short, FACET enables the participants in these groups to engage with their own intervention, amend it and set their own priorities, goals and targets, emphasising prudent health care principles.

Participants in all groups are followed up after 12 weeks. Assessments will be completed face-to-face at the facilities, or at home, dependent upon the participant's needs.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and over
* Willingness to give informed consent, to be randomized to one of the study groups, and comply with all study requirements
* Community dwelling, assisted living conditions or care home residents.
* Ability to walk 10 m independently, or with support if using a cane or walker.
* Ability to understand instructions regarding the use of the technology and execution of the exercise program.

Exclusion Criteria:

* Moderate/severe dementia at baseline (defined as Mini Mental State Examination < 23),
* Severe, disabling stroke at baseline within the previous 6 months (defined as new or previous stroke with Barthel Index < 9),
* Recent (< 3 months prior randomisation) myocardial infarction, or unstable angina.
* Currently undergoing treatment that includes exercise and diet advice by health professionals
* Referred at discharge for condition-specific rehabilitation (e.g. pulmonary rehabilitation, stroke rehabilitation) within the previous 6 months.
* Currently taking part in another study or taken part in an intervention study in the previous six months

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Draper, PhD, Study Director — Aberystwyth University
Locations (1):
- Aberystwyth University, Aberystwyth, Ceredigion, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valdes-Aragones M, Perez-Rodriguez R, Carnicero JA, Moreno-Sanchez PA, Oviedo-Briones M, Villalba-Mora E, Abizanda-Soler P, Rodriguez-Manas L. Effects of Monitoring Frailty Through a Mobile/Web-Based Application and a Sensor Kit to Prevent Functional Decline in Frail and Prefrail Older Adults: FACET (Frailty Care and Well Function) Pilot Randomized Controlled Trial. J Med Internet Res. 2024 Oct 22;26:e58312. doi: 10.2196/58312. PMID 39436684

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done via invitation of existing database from our Research Unit, word of mouth and local advertising and promotion.
Pre-assignment Details: One participant was excluded from the study due to baseline disability status and withdrawal after enrolment is not included in this number. A total of 43 were thus reduced to 42.
  Four participants were re-allocated to 'no online support' arm due to lack of access to internet. One participant was re-allocated to 'Professional led' arm due to not engaging with Patient Empowered activities prior to second visit.
Groups:
- Professional Led With Online Support: The consultation is led by the professional and lifestyle recommendations are based on ViviFrail recommendations and personal experience of the professional.
  The 12-week intervention includes access to an online monitoring platform. The online platform provides the lifestyle recommendations and consists of a diary of activities, examples of exercises, general advice and instructions for monitoring and self-assessment.
  Consultation: The consultation will provide advice (including a short written report) about promoting healthy lifestyles, tailored to the individual
  Online Support: The participant will have access to an online platform 'FACET', to monitor themselves periodically, obtain feedback about their functional ability, receive recommended diet, exercise and physical activity interventions and record the adherence to any intervention.
- Professional Led Without Online Support: The consultation is led by the professional and lifestyle recommendations are based on ViviFrail recommendations and personal experience of the professional.
  There is no access to the online monitoring platform, and lifestyle recommendations were provided on paper to the participant.
  Consultation: The consultation will provide advice (including a short written report) about promoting healthy lifestyles, tailored to the individual
- Patient Empowered With Online Support: The consultation is led by the participant, and started with the questions 'What matters to you', and 'What are your goals'. The professional based the lifestyle recommendations based on these responses.
  The 12-week intervention includes access to an online monitoring platform. The online platform provides the lifestyle recommendations and consists of a diary of activities, examples of exercises, general advice and instructions for monitoring and self-assessment.
  Consultation: The consultation will provide advice (including a short written report) about promoting healthy lifestyles, tailored to the individual
  Online Support: The participant will have access to an online platform 'FACET', to monitor themselves periodically, obtain feedback about their functional ability, receive recommended diet, exercise and physical activity interventions and record the adherence to any intervention.
  Empowered: Actively encouraged to contribute to their own consultation
- Patient Empowered Without Online Support: The consultation is led by the participant, and started with the questions 'What matters to you', and 'What are your goals'. The professional based the lifestyle recommendations based on these responses.
  There is no access to the online monitoring platform, and lifestyle recommendations were provided on paper to the participant.
  Consultation: The consultation will provide advice (including a short written report) about promoting healthy lifestyles, tailored to the individual
  Empowered: The participant will be actively encouraged to contribute to their own consultation and take co-ownership and responsibility for the action plan.
Period: Overall Study
Arm/Group | Professional Led With Online Support | Professional Led Without Online Support | Patient Empowered With Online Support | Patient Empowered Without Online Support
Started | 10 | 11 | 10 | 11
Completed | 10 | 10 | 9 | 11
Not Completed | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Two participants removed as part of the analysis as part of the pilot project. One participant was in Patient Empowered with Online Support (lost to follow up), and another one in Professional led without online support (lost to follow up).
  Another participant was excluded before group allocation due to not meeting the eligibility criteria identified during the pre-enrolment meeting. In total, 43 participants were recruited.
Groups:
- Total: Total of all reporting groups
Arm/Group | Professional Led With Online Support | Professional Led Without Online Support | Patient Empowered With Online Support | Patient Empowered Without Online Support | Total
Number analyzed (Participants) | 10 | 11 | 10 | 11 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 1 | 3
  >=65 years | 9 | 11 | 9 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (6) | 81 (4) | 74 (8) | 75 (6) | 76 (7)
Age, Customized [Count of Participants; unit: Participants]
  60-70 | 2 | 0 | 3 | 1 | 6
  70-80 | 6 | 4 | 3 | 7 | 20
  80-90 | 2 | 7 | 4 | 3 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 9 | 9 | 33
  Male | 3 | 3 | 1 | 2 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 11 | 10 | 11 | 42
Warwick and Edinburgh Mental Well-being Scale [Mean (Standard Deviation); unit: score on a scale] — Score range 14 to 70, with higher scores indicating higher well-being. Population: Incomplete questionnaires were present and excluded from analysis.
  score on a scale
    number analyzed (Participants) | 9 | 8 | 9 | 10 | 36
    (all) | 58 (5) | 55 (5) | 52 (5) | 47 (12) | 53 (9)
Short Physical Performance Battery [Mean (Standard Deviation); unit: score on a scale] — Consists of Walking speed, balance, and chair stand test performance. Scored based on a score of 0-4 on each test, which are summed together. A total maximum score of 12 reflecting good physical performance and better outcomes.
  score on a scale | 11.1 (1.1) | 10.4 (1.5) | 10.7 (1.6) | 10.1 (1.4) | 10.6 (1.4)
SNAQ - Dietary Analysis [Mean (Standard Deviation); unit: units on a scale] — The SNAQ was used to provide a single outcome variable for this. Was originally:
  Food diary and urine metabolomics for the ingestion of food components (meats, fish, legumes and fruits), with emphasis on the quantification of the total protein intake.
  SNAQ: Simplified Nutritional Appetite Questionnaire. Scale from 5-25, with higher scores indicating better outcome Population: Incomplete questionnaires were present and excluded from analysis.
  units on a scale
    number analyzed (Participants) | 10 | 8 | 7 | 10 | 35
    (all) | 15.8 (1.9) | 16.4 (1.8) | 17.1 (0.9) | 16 (2.1) | 16.3 (1.8)
Timed-up-and go [Mean (Standard Deviation); unit: seconds] — The ability to get up from a chair, walk three meters to turn around a cone, and return to sit down again.
  seconds | 7.70 (1.96) | 9.41 (2.86) | 10.98 (9.61) | 10.15 (2.73) | 9.54 (5.01)
Quality of Life SF36 [Mean (Standard Deviation); unit: units on a scale] — the Quality of Life Short Form -36. Scored with the total score (0-100), and higher scores reflecting better quality of life. Population: Incomplete questionnaires were present and excluded from analysis.
  units on a scale
    number analyzed (Participants) | 9 | 8 | 7 | 9 | 33
    (all) | 73 (14) | 66 (19) | 59 (16) | 62 (19) | 66 (17)
Grip Strength [Mean (Standard Deviation); unit: kilogram] — Measured with a hand held grip dynamometer. Measured in kilograms, with higher values reflecting higher strength
  kilogram | 28.6 (4.1) | 24.5 (8.9) | 28.4 (8.9) | 26.8 (9.1) | 27.0 (7.9)
Six Minute Walking Performance [Mean (Standard Deviation); unit: meter] — Quantifies the distance able to walk during six minutes Population: One Participant opted out of completing this task.
  meter
    number analyzed (Participants) | 10 | 9 | 10 | 11 | 40
    (all) | 446 (90) | 393 (96) | 377 (129) | 441 (71) | 416 (99)

OUTCOME MEASURES:

1. Primary Outcome: Pilot Evaluation - Percentage of Participants Retained at Follow up
Description: Percentage of participants returned at follow up, reflects the ability to recruit and retain participants.
  Recruitment took place over a period of 3 months, to recruit 42 participants, with a recruitment rate of 14 participants per month.
Time Frame: 3 Months
Population: A total of 105 people were actively approached, but the project was also promoted via word of mouth and public recruitment interactions and flyers in the local area.
Measure: Count of Participants; unit: Participants
Arm/Group | Professional Led With Online Support | Professional Led Without Online Support | Patient Empowered With Online Support | Patient Empowered Without Online Support
Number analyzed (Participants) | 10 | 11 | 10 | 11
Participants | 10 | 10 | 9 | 11

2. Primary Outcome: Warwick-Edinburgh Mental Well-being Scale (WEMWBS)
Description: Scored with the total score ( range of 14-70), and higher scores reflecting better well-being.
Time Frame: 3 months
Population: Incomplete questionnaires were present and excluded from analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Professional Led With Online Support | Professional Led Without Online Support | Patient Empowered With Online Support | Patient Empowered Without Online Support
Number analyzed (Participants) | 9 | 8 | 9 | 10
score on a scale | 55 (7) | 54 (8) | 53 (7) | 50 (11)
Statistical Analysis 1: Comparison: Professional Led With Online Support vs Professional Led Without Online Support vs Patient Empowered With Online Support vs Patient Empowered Without Online Support; Partial Eta Squared was calculated based on ANOVA with Time (pre-post) as within subject factor and Empowerment (Professional led versus Patient Empowered) as between subject factor; Test type: Superiority; Partial Eta Squared = 0.058

3. Primary Outcome: Short Physical Performance Battery
Description: Consists of Walking speed, balance, and chair stand test performance. Scored based on a score of 0-4 on each test, which are then added. A total maximum score of 12 reflecting good physical performance and thus higher scores indicate better outcome..
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Professional Led With Online Support | Professional Led Without Online Support | Patient Empowered With Online Support | Patient Empowered Without Online Support
Number analyzed (Participants) | 10 | 10 | 9 | 11
score on a scale | 11.4 (1.0) | 10.3 (2.5) | 10.4 (3.0) | 11.1 (1.0)
Statistical Analysis 1: Comparison: Professional Led With Online Support vs Professional Led Without Online Support vs Patient Empowered With Online Support vs Patient Empowered Without Online Support; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Partial Eta Squared = 0.008

4. Secondary Outcome: SNAQ -Dietary Analysis
Description: The SNAQ was used to provide a single outcome variable for this. Was originally:
  Food diary and urine metabolomics for the ingestion of food components (meats, fish, legumes and fruits), with emphasis on the quantification of the total protein intake.
  SNAQ: Simplified Nutritional Appetite Questionnaire. Scale from 5-25, with higher scores indicating better outcome
Time Frame: 3 months
Population: Incomplete questionnaires were present and excluded from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Professional Led With Online Support | Professional Led Without Online Support | Patient Empowered With Online Support | Patient Empowered Without Online Support
Number analyzed (Participants) | 10 | 8 | 7 | 10
units on a scale | 16 (2.1) | 15.6 (2.3) | 17.4 (1.1) | 16.4 (2.4)

5. Secondary Outcome: Timed-up-and go
Description: The ability to get up from a chair, walk three meters to turn around a cone, and return to sit down again.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Professional Led With Online Support | Professional Led Without Online Support | Patient Empowered With Online Support | Patient Empowered Without Online Support
Number analyzed (Participants) | 10 | 10 | 9 | 11
seconds | 7.11 (1.56) | 10.55 (7.04) | 10.00 (9.31) | 8.46 (2.29)

6. Secondary Outcome: Quality of Life SF36
Description: the Quality of Life Short Form -36. Scored with the total score (0-100), and higher scores reflecting better quality of life.
Time Frame: 3 months
Population: Incomplete questionnaires were present and excluded from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Professional Led With Online Support | Professional Led Without Online Support | Patient Empowered With Online Support | Patient Empowered Without Online Support
Number analyzed (Participants) | 9 | 8 | 7 | 9
units on a scale | 72 (21) | 69 (19) | 64 (18) | 60 (19)

7. Secondary Outcome: Grip Strength
Description: Measured with a hand held grip dynamometer. Measured in kilograms, with higher values reflecting higher strength
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Professional Led With Online Support | Professional Led Without Online Support | Patient Empowered With Online Support | Patient Empowered Without Online Support
Number analyzed (Participants) | 10 | 10 | 9 | 11
kilogram | 30.0 (3.7) | 24.7 (7.6) | 28.0 (9.4) | 27.4 (8.1)

8. Other Pre Specified Outcome: Six Minute Walking Performance
Description: Quantifies the distance able to walk during six minutes
Time Frame: 3 months
Population: Some participants opted out of completing the task
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Professional Led With Online Support | Professional Led Without Online Support | Patient Empowered With Online Support | Patient Empowered Without Online Support
Number analyzed (Participants) | 10 | 9 | 9 | 10
meter | 480 (89) | 396 (102) | 407 (163) | 439 (102)

ADVERSE EVENTS:
Time Frame: Three months, the duration of the intervention and the time between baseline and follow up assessment
Arm/Group | Professional Led With Online Support | Professional Led Without Online Support | Patient Empowered With Online Support | Patient Empowered Without Online Support
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 3/11 | 0/10 | 3/11
Other Adverse Events (participants affected / at risk) | 1/10 | 3/11 | 1/10 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Professional Led With Online Support (N=10) | Professional Led Without Online Support (N=11) | Patient Empowered With Online Support (N=10) | Patient Empowered Without Online Support (N=11)
Hernia operation and complications (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant opted for pre-existing hernia to be operated during the intervention period. Caused complications and resulted in hospitalisation. Not deemed to be caused by the intervention.
Progressed into disability and housebound (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant declined in physical functioning and became housebound and was hospitalised. Had severe frailty at baseline and showed extremely low performance scores and was unable to complete most of them, was 'lost to follow up'.
Sepsis and bowel abscess (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant was hospitalised for 6 weeks. Participant indicated it was not related to intervention.
Hip replacement surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant underwent hip replacement surgery during the intervention, from pre-existing condition. Participant deemed it had gotten worse during the intervention
Mental ill-health: stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant was admitted to mental health ward for several weeks and recovered. Participant reported 'over-committed to various activities', of which the intervention was one.
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant spent one night in hospital for observation. Participant deemed it was not related to intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Professional Led With Online Support (N=10) | Professional Led Without Online Support (N=11) | Patient Empowered With Online Support (N=10) | Patient Empowered Without Online Support (N=11)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Fall (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The incomplete data comprised questionnaires that were completed at home and returned subsequently. Adverse events were not recorded by 13 out of 40 participants, but the documentation did not contain a confirmation box to indicate that 'no adverse events' took place. Thus, although it was assumed that these individuals had no adverse events, it is an assumption, based on non-reporting of adverse events and conversations, but not verified in writing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT03707145/Prot_SAP_000.pdf